CLINICAL TRIAL: NCT05751590
Title: Combined Use of Glidescope With Fiber Optic Broncscopy Versus Fiber Optic Alone in Difficult Intubation: a Randomized Clinical Trial
Brief Title: Combined Use of Glidescope With Fiber Optic Broncscopy Versus Fiber Optic Alone in Difficult Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R08/2023
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glidescope + Fiberoptic broncscopy (Active Comparator)
  Interventions: Device: comined use of gliddescope and fiberoptic broncscopy
- Fiberoptic broncscopy (Active Comparator)
  Interventions: Device: fiberoptic bronscopy

INTERVENTIONS:
Device: comined use of gliddescope and fiberoptic broncscopy — endotrachotreal intubation will be done by combined use of Glidescope and Fiberoptic broncscopy
  Arms: Glidescope + Fiberoptic broncscopy
Device: fiberoptic bronscopy — endotrachotreal intubation will be done by Fiberoptic broncscopy
  Arms: Fiberoptic broncscopy

SUMMARY:
In spite of the development of a lot of airway devices in the past 2 decades, tracheal intubation problems were the most common primary airway problems.

The GlideScope® Video Laryngoscope (Verathon, Bothell, WA) is a video laryngoscopy system with a two-segment blade, the distal portion of which houses a charge-coupled device that contains a micro-video camera that transmits images to a 7-inch video liquid crystal display (LCD) monitor. The GlideScope® can be used for routine intubation but is also commonly used as an alternative device for difficult or failed airways. It is particularly useful in cases where cervical motion or mouth opening is limited, preventing creation of a "straight line" of sight from the operator to the glottis .

GlideScope improves the laryngeal view as one of its advantages due to the blade angle of 60° which is designed to improve the glottic view without the need of alignment of the oral, pharyngeal, and tracheal axes and also without adding additional lifting force.

Fibreoptic intubation with a flexible bronchoscope is an important airway management skill in which anaesthesiologists should be proficient. Unfortunately, clinical experience shows that even with reasonable experience and practice, fibreoptic intubation can be challenging. It requires a high degree of manual dexterity, an ability to manoeuvre quickly under stressful clinical situations, and rigorous training and practice to maintain a high level of skill.

Thus, whereas fibreoptic intubatThus, whereas fibreoptic intubation can be used rapidly for intubation, video laryngoscopy may be an effective alternative, especially in patients with an anticipated difficult airway. However, it remains unclear whether video-assisted airway management using the GlideScope provides significant advantages over flexible bronchoscopy in patients with potentially difficult airways , Video laryngoscopy is increasingly used for difficult airway management in anaesthesia, intensive care units and emergency departments. Recently, video laryngoscopy has been incorporated into various difficult airway management algorithms, being recommended as one of the initial steps in the management of difficult airways .

ELIGIBILITY:
Inclusion Criteria:

* patients who will be scheduled for elective surgery requiring orotracheal or nasotracheal intubation with anticipated difficult intubation.
* physical status American Society of Anesthesiologists (ASA) I - III.

Exclusion Criteria:

* Patients who refuse to participate
* patients with body mass index (BMI) >35 kg/m2
* coagulopathy, severe thrombocytopenia <50×103.
* Pregnant females
* physical status American Society of Anesthesiologists (ASA)>IV
* patients requiring rapid sequence induction
* patients with closed mouth opening who are candidates only for nasal intubation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Endotracheal intubation | 1st seconds till succesfull intubation
  Intubation time is defined as the time from insertion of either the GlideScope combined with the Fiberoptic broncscopy or the Fiberoptic broncscopy alone into the mouth, to the time when end tidal CO2 exceeded (20 mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt